CLINICAL TRIAL: NCT03137433
Title: Enhancing Weight Loss With Meal-Replacement Therapy in Teens With Severe Obesity
Brief Title: Weight Loss With Meal-Replacement Therapy in Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2017-25609
Record Dates: First submitted 2017-04-25; First posted 2017-05-02 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Severe; Pediatric Obesity
Keywords: Weight loss; Cardiometabolic; Meal-replacement therapy
MeSH Terms: conditions — Obesity, Morbid; Pediatric Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal-Replacements (Experimental): Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data).
  Interventions: Dietary Supplement: Meal-replacement Therapy
- Meal-Replacements Plus (Experimental): Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data). This group will be provided additional information to go along with meal-replacements.
  Interventions: Dietary Supplement: Meal-replacement Therapy

INTERVENTIONS:
Dietary Supplement: Meal-replacement Therapy — We seek to examine the effect of meal-replacement therapy on weight loss outcomes in teens with severe obesity.

SUMMARY:
This study seeks to examine whether meal-replacement therapy is able to enhance weight loss among teens with severe obesity. In addition, we are also interested in examining the degree of weight loss needed to improve important cardiometabolic risk factors among adolescents.

DETAILED DESCRIPTION:
This study will involve 130 adolescents (ages 13-17 years old) participating in meal replacement therapy and will last one year (12 months).

Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data). Shakes/meals will be provided free of charge - fruits/vegetables will be purchased by the participants. Guidance will be provided regarding the use of the meal replacement shakes at school, and participants will be encouraged to engage in family meal sessions despite eating different foods.

We will measure the changes in resting metabolic rate, traditional clinical risk markers (TG, HDL-c, LDL-c, TC, glucose, insulin), vascular function, weight-related quality of life, and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥1.2 times the 95th percentile (based on sex and age) or BMI ≥35 kg/m2
* 13-17 years old

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Previous (within 6 months) or current use of meal replacements
* Previous (within 6 months) or current use of medication(s) prescribed primarily for weight loss (refer to appendix material for comprehensive list)
* If currently using weight altering drug(s) for non-obesity indication(s) (refer to appendix material for comprehensive list), any change in drug(s) or dose within the previous 6 months
* Previous bariatric surgery
* If currently using anti-hypertensive medication(s), lipid medication(s), and/or medication(s) to treat insulin resistance (refer to appendix material for comprehensive list), any change in drug(s) or dose within the previous 6 months
* If currently using CPAP/BIPAP (for sleep apnea), change in frequency of use or settings within the previous 6 months
* History of treatment with growth hormone
* Neurodevelopmental disorder severe enough to impair ability to comply with study protocol
* Clinical diagnosis of bipolar illness, schizophrenia, conduct disorder, and/or substance use/abuse
* Females: currently pregnant or planning to become pregnant
* Tobacco use
* Bulimia nervosa
* Endorsement of vomiting, laxative use, and/or diuretic use for weight control (EDE-Q)
* Binge eating disorder
* Neurological disorder
* Hypothalamic obesity
* Obesity associated with genetic disorder (monogenetic obesity)
* Hyperthyroidism or uncontrolled hypothyroidism
* History of cholelithiasis

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Kelly, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gross AC, Freese RL, Bensignor MO, Bomberg EM, Dengel DR, Fox CK, Rudser KD, Ryder JR, Bramante CT, Raatz S, Lim F, Hur C, Kelly AS. Financial Incentives and Treatment Outcomes in Adolescents With Severe Obesity: A Randomized Clinical Trial. JAMA Pediatr. 2024 Aug 1;178(8):753-762. doi: 10.1001/jamapediatrics.2024.1701. PMID 38884967

RESULTS

PARTICIPANT FLOW:
Groups:
- Meal-Replacements Plus: Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data). This group will be provided additional information to go along with meal-replacements; this group of individuals received financial incentives as part of their weight loss.
  Meal-replacement Therapy: We seek to examine the effect of meal-replacement therapy on weight loss outcomes in teens with severe obesity.
Period: Overall Study
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Started | 63 | 63
Completed | 44 | 45
Not Completed | 19 | 18
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 5 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Moved out of study area | 1 | 0
Not completed — Too far out of window due to COVID | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants randomized to each arm at the Baseline visit.
Groups:
- Meal-Replacements Plus: Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data). This group was provided additional information to go along with meal-replacements which was that they would be paid for their weight loss.
  Meal-replacement Therapy: We seek to examine the effect of meal-replacement therapy on weight loss outcomes in teens with severe obesity.
- Total: Total of all reporting groups
Arm/Group | Meal-Replacements | Meal-Replacements Plus | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Categorical [Count of Participants; unit: Participants] — Age at study entry
  Participants
    <=18 years | 63 | 63 | 126
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 28 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 57 | 55 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 43 | 40 | 83
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (From Baseline to 1-year)
Description: Percent change in body mass index (BMI) from baseline to 1-year (kg/m2)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: Percent change in BMI
Groups:
- Meal-Replacements Plus: Participants will be asked to strictly follow the individually-prescribed eating regimen, which will include shakes (breakfast and lunch) and pre-packaged frozen entrée meals for dinner, two servings of fruit, and three servings of vegetables per day. Daily caloric allotment will be tailored for each individual (number of shakes and frozen meals) by calculating the average daily caloric deficit necessary to achieve negative energy balance (using the metabolic rate/energy expenditure data). This group will be provided additional information to go along with meal-replacements, which was a financial incentive for weight loss.
  Meal-replacement Therapy: We seek to examine the effect of meal-replacement therapy on weight loss outcomes in teens with severe obesity.
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
Percent change in BMI | -0.9 (1.3) | -6.6 (1.6)

2. Secondary Outcome: Total Fat Mass (kg)
Description: Change in fat mass from randomization to week 52
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
Kg | -1.3 (1.5) | -6.1 (1.5)

3. Secondary Outcome: Carotid-radial Pulse Wave Velocity (m/s)
Description: Change in measure of arterial stiffness (from baseline to 1-year)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
m/s | -0.1 (0.1) | 0.1 (0.2)

4. Secondary Outcome: Impact of Weight-related on Quality of Life
Description: Impact of Weight-related on Quality of Life Total Transformed Score (from physical comfort transformed score, body self esteem transformed score, social life transformed score, and family relations transformed score). Scores range from 0 to 100 with 100 representing the best quality of life.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
score on a scale | 3.2 (2.5) | 5.2 (3.1)

5. Secondary Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure (from baseline to 1-year)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mm Hg | -3.1 (1.7) | -2.1 (1.7)

6. Secondary Outcome: Diastolic Blood Pressure
Description: Change in diastolic blood pressure (from baseline to 1-year)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mm Hg | -0.3 (1.4) | 0.1 (1.5)

7. Secondary Outcome: Total Cholesterol
Description: Total cholesterol (mg/dL)
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mg/dL | 153.9 (30) | 158.6 (32)

8. Secondary Outcome: HDL
Description: High Density Lipoprotein (mg/dL)
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mg/dL | 43.6 (9) | 44.0 (10)

9. Secondary Outcome: LDL
Description: Low Density Lipoprotein (mg/dL)
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mg/dL | 89.1 (29) | 89.3 (30)

10. Secondary Outcome: Triglyceride/HDL Cholesterol Ratio
Description: Triglyceride/HDL cholesterol ratio (from baseline to 1-year)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: TG/HDL cholesterol ratio
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
TG/HDL cholesterol ratio | -0.2 (0.3) | -0.5 (0.3)

11. Secondary Outcome: Total Glucose
Description: Total Glucose (mg/dL)
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mg/dL | 87.3 (9) | 87.4 (6)

12. Secondary Outcome: Insulin
Description: Insulin (mU/dL)
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mU/dL
Arm/Group | Meal-Replacements | Meal-Replacements Plus
Number analyzed (Participants) | 63 | 63
mU/dL | 28.3 (16) | 34.2 (25)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Meal-Replacements | Meal-Replacements Plus
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/63 | 1/63
Other Adverse Events (participants affected / at risk) | 9/63 | 6/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meal-Replacements (N=63) | Meal-Replacements Plus (N=63)
Exacerbation of Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 — Hospitalization for asthma. Asthma was noted as a pre-existing condition at enrollment.
Suicide attempt (Psychiatric disorders) | 1 (1) | 0
Overdose (Psychiatric disorders) | 1 (1) | 0
Acquired pneumonia and E-cigarette associated lung injury (EVALI) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meal-Replacements (N=63) | Meal-Replacements Plus (N=63)
Self report of taking laxatives (Psychiatric disorders) | 7 (7) | 6 (9) — Taken from the Eating Disorder Examination-Questionnaire (EDEQ) question 17
Self induced vomiting (Psychiatric disorders) | 9 (10) | 6 (10) — Self report of making oneself sick based on the Eating Disorder Examination-Questionnaire, question 16.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03137433/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03137433/ICF_001.pdf